CLINICAL TRIAL: NCT02370316
Title: Neuroimaging and Clinical Markers of Change in Borderline Personality Disorder After Metacognitive Interpersonal Therapy - Standard Approach
Brief Title: Biomarkers of Change in BPD After Metacognitive Interpersonal Therapy-standard Approach
Acronym: CLIMAMITHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Roberta Rossi, psyD, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR-2011-02351347
Record Dates: First submitted 2015-02-10; First posted 2015-02-24 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Borderline Personality Disorder
Keywords: metacognition; MRI; Psychotherapy
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIT - SA (Experimental): Metacognitive Interpersonal Therapy -standard approach (MIT-SA) is a cognitive behavior-based psychotherapeutic approach that works to increase metacognitive abilities and to improve interpersonal relationships
  Interventions: Behavioral: Metacognitive Interpersonal Therapy (MIT-SA)
- Clinical Structured Treatment (CST) (Active Comparator): Clinical Structured Treatment (CST) is a structured case management and symptom-targeted medication
  Interventions: Behavioral: Clinical Structured Treatment

INTERVENTIONS:
Behavioral: Metacognitive Interpersonal Therapy (MIT-SA) — MIT-SA consists of weekly individual therapy (1 year) and weekly group sessions (six months)
  Arms: MIT - SA
Behavioral: Clinical Structured Treatment — structured case management and symptom-targeted medication
  Arms: Clinical Structured Treatment (CST)

SUMMARY:
The present randomised clinical trial aims to assess the clinical and neurobiological changes following Metacognitive Interpersonal Therapy -standard approach (MIT-SA) compared with Clinical Structured Treatment (CST) derived from specific recommendations in APA guidelines for borderline personality disorder (BPD). The investigators will assess clinical changes in metacognitive abilities and in emotion regulation and changes in brain activation patterns at the resting state and while they view emotional pictures. A multidimensional assessment will be performed at the baseline, at 6, 12, 18 months. The investigators will take structural and functional Magnetic Resonance Images (MRIs) in MIT-Treated BPD (N=30) and CST-treated BPD (N=30) at baseline and after treatment, as well as a group of 30 healthy and unrelated volunteers that will be scanned once for comparison. Furthermore, blood analyses will be done in order to assess level of BDNF and some hormone levels (oxytocin and vasopressin) before and after treatments.

DETAILED DESCRIPTION:
Patients will be randomly allocate to two kind of interventions: MIT-SA and CST. Patients will be enrolled in 3 centres: Unit of Psychiatry, IRCCS San Giovanni di Dio-FBF, Brescia; Terzo Centro di Psicoterapia Cognitiva-School of Cognitive Psychotherapy, Rome; Mental Health Department ASL Roma G, Rome, Italy.

A multidimensional evaluation with standardized tools will assess: level of psychopathology, depression, anger, impulsiveness, level of functioning. In particular, the assessment will include: the Structured Clinical Interview for DSM disorder; the Difficulties in Emotion Regulation Scale (DERS) (primary outcome); Metacognition Assessment Interview to assess metacognitive functions. Neuropsychological assessment will assess different cognitive domains, empathy and emotional recognition with standardized tools . Additionally, the emotional priming paradigm to evaluate emotion processing will be included.

Data on demographics, traumatic exposure, suicide attempts, self-injury and aggression episodes, hospitalizations, and pharmacotherapy will be collected. Structural and functional MRI will be collected in MIT-Treated BPD (N=30) and CST-treated BPD (N=30) at baseline and after treatment. Healthy volunteers (N=30) will be scanned once for comparison. Specific MRI analyses:1) Whole brain (cortical thickness) analyses will be conducted to explore the correlates of psychotherapy and treatment response. Functional connectivity studies will consider A) activity at rest, both before and after treatment; B) functional activation in response to standardized emotional material from the International Affective Pictures System (IAPS). 2) Region of interest analyses: regions of particular elevance (hippocampus, amygdale, insula) will be studied using advanced neuroimaging tools.

Blood samples will be collected in order to assess variations in levels of BDNF and some hormones (oxytocin and vasopressin) pre- and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM 5 criteria for BPD
* Able to provide informed consent

Exclusion Criteria:

* lifetime diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, organic mental syndromes;
* active substance abuse or dependence in the 6 months before the enrolment;
* concurrent psychotherapy;
* cognitive impairment or dementia;
* relevant neurological signs;
* pregnancy/lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Change in Difficulties in Emotion Regulation Scale (DERS) | 6, 12, 18 months
  Clinical changes in metacognitive abilities and in emotion regulation assessed with the Difficulties in Emotion Regulation Scale (DERS)

SECONDARY OUTCOMES:
changes in metacognitive abilities (assessed with the Metacognition Assessment Interview) | 6, 12, 18 months
  Clinical changes in metacognitive abilities assessed with the Metacognition Assessment Interview
Change from Baseline in activation in the amygdala at 12 months | 12 months
  Change from Baseline in activation in the amygdala at 12 months in response to standardized emotional material from the International Affective Pictures System

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Rossi, PsyD, Principal Investigator — IRCCS Centro San Giovanni di Dio - FBF
Locations (1):
- Irccs Centre San Giovanni di Dio - Fatebenefratelli, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Semerari A, Cucchi M, Dimaggio G, Cavadini D, Carcione A, Battelli V, Nicolo G, Pedone R, Siccardi T, D'Angerio S, Ronchi P, Maffei C, Smeraldi E. The development of the Metacognition Assessment interview: instrument description, factor structure and reliability in a non-clinical sample. Psychiatry Res. 2012 Dec 30;200(2-3):890-5. doi: 10.1016/j.psychres.2012.07.015. Epub 2012 Aug 18. PMID 22906953
- [Background] Rossi R, Lanfredi M, Pievani M, Boccardi M, Rasser PE, Thompson PM, Cavedo E, Cotelli M, Rosini S, Beneduce R, Bignotti S, Magni LR, Rillosi L, Magnaldi S, Cobelli M, Rossi G, Frisoni GB. Abnormalities in cortical gray matter density in borderline personality disorder. Eur Psychiatry. 2015 Feb;30(2):221-7. doi: 10.1016/j.eurpsy.2014.11.009. Epub 2015 Jan 2. PMID 25561291
- [Background] Rossi R, Pievani M, Lorenzi M, Boccardi M, Beneduce R, Bignotti S, Borsci G, Cotelli M, Giannakopoulos P, Magni LR, Rillosi L, Rosini S, Rossi G, Frisoni GB. Structural brain features of borderline personality and bipolar disorders. Psychiatry Res. 2013 Aug 30;213(2):83-91. doi: 10.1016/j.pscychresns.2012.07.002. Epub 2012 Nov 10. PMID 23146251
- [Background] Rossi R, Lanfredi M, Pievani M, Boccardi M, Beneduce R, Rillosi L, Giannakopoulos P, Thompson PM, Rossi G, Frisoni GB. Volumetric and topographic differences in hippocampal subdivisions in borderline personality and bipolar disorders. Psychiatry Res. 2012 Aug-Sep;203(2-3):132-8. doi: 10.1016/j.pscychresns.2011.12.004. Epub 2012 Sep 1. PMID 22944368
- [Derived] Quattrini G, Carcione A, Lanfredi M, Nicolo G, Pedrini L, Corbo D, Magni LR, Geviti A, Ferrari C, Gasparotti R, Semerari A, Pievani M, Rossi R. Effect of metacognitive interpersonal therapy on brain structural connectivity in borderline personality disorder: Results from the CLIMAMITHE randomized clinical trial. J Affect Disord. 2025 Jan 15;369:1145-1152. doi: 10.1016/j.jad.2024.10.107. Epub 2024 Oct 23. PMID 39454963
- [Derived] Rossi R, Corbo D, Magni LR, Pievani M, Nicolo G, Semerari A, Quattrini G, Riccardi I, Colle L, Conti L, Gasparotti R, Macis A, Ferrari C, Carcione A; CLIMAMITHE study group. Metacognitive interpersonal therapy in borderline personality disorder: Clinical and neuroimaging outcomes from the CLIMAMITHE study-A randomized clinical trial. Personal Disord. 2023 Jul;14(4):452-466. doi: 10.1037/per0000621. Epub 2023 May 25. PMID 37227866
- [Derived] Magni LR, Carcione A, Ferrari C, Semerari A, Riccardi I, Nicolo' G, Lanfredi M, Pedrini L, Cotelli M, Bocchio L, Pievani M, Gasparotti R, Rossi R; CLIMAMITHE Study group. Neurobiological and clinical effect of metacognitive interpersonal therapy vs structured clinical model: study protocol for a randomized controlled trial. BMC Psychiatry. 2019 Jun 24;19(1):195. doi: 10.1186/s12888-019-2127-2. PMID 31234864